CLINICAL TRIAL: NCT04657861
Title: Clinical Trial for the Safety and Efficacy of APRIL CAR-T Cells Therapy for Patients With BCMA/TACI Positive Relapsed and/or Refractory Multiple Myeloma
Brief Title: APRIL CAR-T Cell Therapy for Patients With BCMA/TACI Positive Relapsed and/or Refractory Multiple Myeloma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APRIL-001
Record Dates: First submitted 2020-10-22; First posted 2020-12-08 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-03

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma, Refractory
Keywords: Multiple Myeloma; CAR T-cell therapy; BCMA/TACI positive
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of APRIL CAR T-cells (Experimental): Each subject receive APRIL CAR T-cells by intravenous infusion
  Interventions: Drug: APRIL CAR-T cells

INTERVENTIONS:
Drug: APRIL CAR-T cells — Each subject receive APRIL CAR T-cells by intravenous infusion
  Other Names: APRIL CAR-T cells injection

SUMMARY:
A study of APRIL CAR-T cells therapy for patients with BCMA/TACI positive relapsed and/or refractory multiple myeloma

DETAILED DESCRIPTION:
This is a single arm, open-label, single-center study. This study is indicated for relapsed or refractory BCMA/TACI positive relapsed and/or refractory multiple myeloma. The selections of dose levels and the number of subjects are based on clinical trials of similar foreign products. 36 patients will be enrolled. Primary objective is to explore the safety, main consideration is dose-related safety.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of BCMA/TACI+ multiple myeloma (MM)：

   1. Patients with MM relapsed after BCMA CAR-T therapy; Or MM with positive BCMA/TACI expression;
   2. Relapsed after hematopoietic stem cell transplantation;
   3. Cases with recurrent positive minimal residual disease;
   4. Extramedullary leision which is hard to be eradicated by chemotherapy or radiotherapy.
2. Male or female aged 18-75 years;
3. Total bilirubin ≤ 51 umol/L, ALT and AST ≤ 3 times of upper limit of normal, creatinine ≤ 176.8 umol/L;
4. Echocardiogram shows left ventricular ejection fraction (LVEF) ≥50%;
5. No active infection in the lungs, blood oxygen saturation in indoorair is ≥ 92%;
6. Estimated survival time ≥ 3 months;
7. ECOG performance status 0 to 2;
8. Patients or their legal guardians volunteer to participate in the studyand sign the informed consent.

Exclusion Criteria:

Subjects with any of the following exclusion criteria were not eligible for this trial:

1. History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular, hemorrhagic diseases;
2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
3. Pregnant (or lactating) women;
4. Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis);
5. Active infection of hepatitis B virus or hepatitis C virus;
6. Concurrent therapy with systemic steroids within 2 weeks prior to screening, except for the patients recently or currently receiving in haled steroids;
7. Previously treated with any CAR-T cell product or other genetically modified T cell therapies;
8. Creatinine>2.5mg/dl, or ALT / AST > 3 times of normal amounts, or bilirubin>2.0 mg/dl;
9. Other uncontrolled diseases that were not suitable for this trial;
10. Patients with HIV infection;
11. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2024-08-20 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after APRIL targeted CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Time Frame: Up to 2 years after APRIL targeted CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Multiple Myeloma (MM), Overall response rate (ORR) | At Month 1, 3, 6, 12, 18 and 24
  Assessment of ORR (ORR = sCR+CR+VGPR+PR+MR) at Month 1, 3, 6, 12, 18 and 24
MM, Overall survival (OS) | Up to 2 years after APRIL CAR-T cells infusion
  From the first infusion of APRIL CAR-T cells to death or the last visit
MM, Event-free survival (EFS) | Up to 2 years after APRIL CAR-T cells infusion
  From the first infusion of APRIL CAR-T cells to the occurrence of any event, including death, relapse or gene relapse, disease progression (any one occurs first), and the last visit
Quality of life including sports activity | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) scale [For item1-28: max score: 112, min score: 28, higher scores mean a better outcome; for item 28-29: max score: 14, min score: 2, higher scores mean a worse outcome] to measure Quality of life at Baseline, Month 1, 3, 6, 9 and 12
Activities of Daily Living (ADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Activities of Daily Living (ADL) scale (Barthel Index) [max score: 100, min score: 0, higher scores mean a better outcome] at Baseline, Month 1, 3, 6, 9 and 12
Instrumental Activities of Daily Living (IADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment of Instrumental Activities of Daily Living (IADL) scale [max score: 56, min score: 14, higher scores mean a worse outcome] at Baseline, Month 1, 3, 6, 9 and 12
Hospital Anxiety and Depression Scale (HADS) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Hospital Anxiety and Depression Scale (HADS) [max score: 42, min score: 0, higher scores mean a worse outcome] at Baseline, Month 1, 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital，College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No